CLINICAL TRIAL: NCT04809987
Title: Evaluation of Effectiveness of Virtual Gait System Intervention in Motor Function, Tone and Sensibility, in People with Incomplete Spinal Cord Injury.
Brief Title: Effectiveness of Virtual Gait System Intervention in Motor Function in People with Incomplete Spinal Cord Injury.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Pilar Serra Añó, Chaired Full Professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09102019
Record Dates: First submitted 2020-12-01; First posted 2021-03-22 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Incomplete Spinal Cord Injury
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Virtual Gait and Physical Exercise (Experimental)
  Interventions: Other: Virtual Gait; Other: Physical Exercise
- Documental projection and Physical Exercise (Sham Comparator)
  Interventions: Other: Physical Exercise; Other: Documental projection
- Virtual Gait (Experimental)
  Interventions: Other: Virtual Gait
- Documental Projection (Sham Comparator)
  Interventions: Other: Documental projection

INTERVENTIONS:
Other: Virtual Gait — The subject will be stand up with a standing opposite a mirror (from the waist up) and a screen (from the waist down) where a video of treadmill gait of a person will be projected.
  Arms: Virtual Gait; Virtual Gait and Physical Exercise
Other: Physical Exercise — Specific gait exercise was conducted.
  Arms: Documental projection and Physical Exercise; Virtual Gait and Physical Exercise
Other: Documental projection — The subject will be stand up with a standing opposite a mirror (from the waist up) and a screen (from the waist down) where video without any type of animal or human movement was showed.
  Arms: Documental Projection; Documental projection and Physical Exercise

SUMMARY:
Roughly 60% of people with Spinal Cord Injury (SCI) have an incomplete one, with a strength, sensibility, and muscle tone alteration. Moreover, this condition involves a high impact on the psychological and socioeconomic levels.

After an incomplete SCI, spontaneous functional recovery occurs. This recovery is strong associated with injury and person characteristics, and with corticospinal fibers, motor cortex, and spinal neurons neuroplasticity. However, also it is possible to stimulate neuroplasticity mechanisms of these structures throughout rehabilitation techniques. Generally, with external devices, exoskeletons, or physical exercise therapy. With it, clinicians achieve early, intensive and specific therapies.

This reorganization and recovery can be influenced because of mirror neurons, located in motor and premotor areas, and in other cortical and subcortical areas. These types of neurons are activated with a functional action observation.

Due to incomplete SCI neuroplasticity recover, these therapies (concretely, illusion visual systems) have been the object of systematic review in this population with the aim of knowing its repercussion on neuropathic pain in chronic patients. Moseley and collaborators in 2007 were the first of proposing a virtual gat system that induced patients' gait illusion. The promising results in this intervention, leading institutions performed similar studies with other stimuli and devices, with good results.

However, SCI studies are focused on neuropathic pain and not in motor function (like in other populations). Therefore, there is not any study that assesses mirror neurons activity in the physical condition and/or in functional gait capaity in incomplete spinal cord injury population.

On the basis of the above, the study principal aim is to evaluate a virtual gait treatment effectiveness compared with combined interventions with specific gait physical exercise in functional capacity in the incomplete spinal cord injury population. Concretely in follow outcomes: gait, functionality, strength, muscle tone, sensibility, and neuropathic pain.

DETAILED DESCRIPTION:
Roughly 60% of people with Spinal Cord Injury (SCI) have an incomplete one, with a strength, sensibility, and muscle tone alteration. Moreover, this condition involves a high impact on the psychological and socioeconomic levels.

After an incomplete SCI, spontaneous functional recovery occurs. This recovery is strong associated with injury and person characteristics, and with corticospinal fibers, motor cortex, and spinal neurons neuroplasticity. However, also it is possible to stimulate neuroplasticity mechanisms of these structures throughout rehabilitation techniques. Generally, with external devices, exoskeletons, or physical exercise therapy. With it, clinicians achieve early, intensive and specific therapies.

This reorganization and recovery can be influenced because of mirror neurons, located in motor and premotor areas, and in other cortical and subcortical areas. These types of neurons are activated with a functional action observation. Mirror neurons activity has been studied with several brain injury populations (Cranial traumatisms, Parkinson, or Alzheimer's disease). Therefore, several experimental investigations have been developed by applying different interventions to modified their activity (mirror therapies, virtual reality therapies, or Action-Observation therapies). Its results showed promising improvements, except for advanced Alzheimer's disease.

Due to incomplete SCI neuroplasticity recover, these therapies (concretely, illusion visual systems) have been the object of systematic review in this population with the aim of knowing its repercussion on neuropathic pain in chronic patients. Moseley and collaborators in 2007 were the first of proposing a virtual gat system that induced patients' gait illusion. The promising results in this intervention, leading institutions performed similar studies with other stimuli and devices, with good results.

However, SCI studies are focused on neuropathic pain and not in motor function (like in other populations). Therefore, there is not any study that assesses mirror neurons activity in the physical condition and/or in functional gait capaity in incomplete spinal cord injury population.

On the basis of the above, the study principal aim is to evaluate a virtual gait treatment effectiveness compared with combined interventions with specific gait physical exercise in functional capacity in the incomplete spinal cord injury population. Concretely in follow outcomes: gait, functionality, strength, muscle tone, sensibility, and neuropathic pain.

Therefore, this study is a randomized clinical trial in which four groups of twenty people in each group will participate, with different interventions:

1. Virtual Gait and Physical exercise.
2. Documental projection and physical exercise.
3. Virtual Gait.
4. Documental Projection.

Data analysis will be performed with SPSS statistic program (v26). Normality and homocedasticity will be analyzed by Shapiro-Wilk t-test and Levene test, respectively. For comparation between groups Bonferroni will be used. If any confusion factor that not meet requirements to be analysed like a covaraible exist, ANCOVA will be used. When p<0.0.5 statistical significant differences will be asumed.

ELIGIBILITY:
Inclusion Criteria:

* Incomplete spinal cord injury (ASIA C,D or E).
* Mini-Mental State Examination >23 points.

Exclusion Criteria:

* Lower limbs traumathic pathology.
* Other nervous system alterations.
* Vestibular diseases.
* Other diseases.

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-01-30 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Gait | 10 minutes
  10 meters Walking Test
Functionality | 10 minutes
  FallSkip
Strength | 10 minutes
  Load Cell

SECONDARY OUTCOMES:
Spasticity | 10 minutes
  MyotonPRO
Neuropathic Pain | 10 minutes
  Brief Pain Inventory
Muscle Activation | 10 minutes
  EMG

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Faculty of Physiotherapy, Valencia, Spain
  - Facultat de Fisioterapia, Universitat de València, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Moseley LG. Using visual illusion to reduce at-level neuropathic pain in paraplegia. Pain. 2007 Aug;130(3):294-298. doi: 10.1016/j.pain.2007.01.007. Epub 2007 Mar 1. PMID 17335974
- [Derived] Molla-Casanova S, Munoz-Gomez E, Moreno-Segura N, Ingles M, Aguilar-Rodriguez M, Sempere-Rubio N, Serra-Ano P. Effect of a virtual walking and exercise-based intervention on muscle strength and activation in people with incomplete spinal cord injury. Sci Rep. 2025 Jan 24;15(1):3144. doi: 10.1038/s41598-025-86845-8. PMID 39856165